CLINICAL TRIAL: NCT03698773
Title: Satisfaction of Pain Relief During Labor and Delivery Following Access to New Educational Materials
Brief Title: Pain Relief Satisfaction With New Educational Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Kathleen Reyes, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 18-642
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Results first posted 2024-06-24 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Group (Active Comparator): Access to existing educational materials about labor/delivery pain relief options, as well as an opportunity to ask physicians, nurses, and other relevant personnel for more information.
  Interventions: Other: Access to routine information
- Website Group (Experimental): Access to a tablet computer set to display an educational website (thepainlesspush.com) with information about labor/delivery pain relief options, as well as an opportunity to ask physicians, nurses, and other relevant personnel for more information.
  Interventions: Other: Access to website

INTERVENTIONS:
Other: Access to routine information — Access to routine pain-control information
  Arms: Baseline Group
Other: Access to website — Access to informational website: thepainlesspush.com
  Arms: Website Group

SUMMARY:
This study compares patient satisfaction after labor and delivery with access to either the default educational materials available, or to a table computer set to display an educational website, thepainlesspush.com.

DETAILED DESCRIPTION:
This is a prospective randomized controlled study. The investigators hypothesize that parturients with access to the website will exhibit greater satisfaction with labor and delivery pain control.

Potential participants will be recruited from the University of New Mexico Hospital (UNMH) Labor & Delivery floor. Patients will be enrolled following an oral consent process. They will be randomized into either control group or intervention group. Control group participants will have their standard of care visit with an anesthesiologist and routine hospital pain-relief information. Intervention group participants will have their standard of care visit with an anesthesiologist, plus one hour in which to view the patient education website thepainlesspush.com, on an iPad provided by the Anesthesiology department for this purpose. After their delivery and transfer to the mother/baby unit, participants will complete a satisfaction survey brought to them by a study team member. Participants will complete the survey following their delivery and prior to discharge. The primary team will notify us with expected discharge in which we will retrieve the survey from them in their room and answer any last questions. Their active participation in the study will be complete at this time. After a participant completes the satisfaction survey, research team members will collect demographic information and relevant obstetric/medical history information from the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* All English- or Spanish-speaking patients who are admitted to UNMH Labor and Delivery for planned progression to active labor.

Exclusion Criteria:

* Age under 18 years
* Patients unable to provide consent for medical procedures
* Patients who do not speak either English or Spanish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Reyes, MD, Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Baseline Group | Website Group
Started | 50 | 56
Completed | 48 | 55
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Group | Website Group | Total
Number analyzed (Participants) | 50 | 56 | 106
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 28 [25 to 32] | 29 [25 to 32] | 29 [25 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 56 | 106
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 56 | 106
Language preference [Count of Participants; unit: Participants]
  English | 39 | 43 | 82
  Spanish | 9 | 12 | 21
  Unknown | 2 | 1 | 3
Had chosen preferred labor analgesia type before hospital arrival [Count of Participants; unit: Participants] — Count of participants who had chosen a preferred type of labor analgesia during pregnancy, before arriving at the hospital for labor
  Participants | 40 | 42 | 82
Arrived at hospital desiring labor epidural [Count of Participants; unit: Participants] — Count of participants who had chosen labor epidural as the preferred type of analgesia during pregnancy, before arriving at the hospital for labor
  Participants | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction With Pain Control in Labor
Description: Satisfaction as measured by agreement with Likert scale questionnaire item "I was satisfied with my choice for pain control in labor" where 1 = strongly disagree, 3 = neither agree nor disagree, and 5 = strongly agree. High scores indicate high satisfaction.
Time Frame: Following delivery and prior to discharge, up to two days
Population: Data on this outcome are available for n=97 participants total. A total of 9 participants (4 in the Baseline group and 5 in the Website group) did not provide data on the primary outcome.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Baseline Group | Website Group
Number analyzed (Participants) | 46 | 51
score on a scale | 5 [3 to 5] | 5 [4 to 5]
Statistical Analysis 1: Comparison: Baseline Group vs Website Group; Test type: Superiority; p = 0.16, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Epidural Analgesia Utilization Rate
Description: Number of patients receiving epidural analgesia
Time Frame: On day of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Group | Website Group
Number analyzed (Participants) | 48 | 55
Participants | 41 | 46
Statistical Analysis 1: Comparison: Baseline Group vs Website Group; Test type: Superiority; p > 0.99, Fisher Exact

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | Baseline Group | Website Group
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/43
Other Adverse Events (participants affected / at risk) | 0/37 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03698773/Prot_SAP_000.pdf